CLINICAL TRIAL: NCT05420792
Title: The Effect of Interpersonal Relationships and Social Rhythm Therapy on Biological Rhythm and Relapses in Individuals With Bipolar Disorder
Brief Title: The Effect of Interpersonal Relationships and Social Rhythm Therapy Individuals With Bipolar Disorder
Acronym: IPSRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Yeliz Aktas, PhD Student, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Ege University Nursing
Record Dates: First submitted 2022-06-06; First posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Bipolar Disorder; Bipolar I Disorder; Bipolar II Disorder
Keywords: bipolar disorder; Interpersonal and Social Rhythm Therapy; psychiatric nursing
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): Peplau Interpersonal Relations based IPSRT will be applied to the intervention group
  Interventions: Behavioral: Peplau Interpersonal Relations based IPSRT will be applied to the intervention group
- control group (No Intervention): the control group will be given a Community Mental Health Center and will also continue the treatment

INTERVENTIONS:
Behavioral: Peplau Interpersonal Relations based IPSRT will be applied to the intervention group — IPSRT based on peplau Interpersonal Relations theory will be applied to the intervention group. First of all, information about the study will be given. An informed consent form will be filled and a history will be taken from the patient. With the Life Events Chart, past attacks and life events, interpersonal relations will be compared. Interpersonal Circle will be made to better understand the individual and relationships. A Joint Study Plan, which summarizes the disease history, life events, and interpersonal circle, will be created and presented to the patient in summary form. The patient will be given psychoeducation about his illness, drugs and social rhythms. A Social Rhythm Metric (SRM) will be created and monitored throughout therapy to assess their daily routine. Early warning signs of impending attacks will be discussed, managing symptoms, situations that may disrupt social rhythm will be determined (travel, vacation, moving, changing job)
  Arms: intervention group

SUMMARY:
Interpersonal and Social Rhythm Therapy (IPSRT) is a type of psychotherapy that applies social rhythm theories in bipolar disorder. The purpose of IPSRT is to stabilize people's social routines (daily routines, sleep-wake balances), gain insight into the two-way relationship between interpersonal events and mood, and increase their satisfaction with social roles.

This study was planned as a follow-up study in a quantitative, randomized controlled experimental design, aiming to determine the effectiveness of Peplau's Interpersonal Relations theory-based IPSRT applied to individuals with bipolar disorder to determine the effect on biological rhythm, interpersonal relationships and relapse frequencies. Pre-intervention pre-test, post-intervention post-test and follow-up scheme will be used. To carrying out of this study, first of all, intervention and control groups will be formed by randomization according to gender and bipolar type (I-II), using the Introductory Information Form, Young Mania Rating and Hamilton Depression Rating Scales from individuals with bipolar disorder registered to the Community Mental Health Service (CMHS). As a pre-test (Introductory Information Form, Young Mania Rating Scale, Hamilton Depression Rating Scale, Biological Rhythm Assessment Interview, Interpersonal Competence Scale) to the intervention and control groups, Peplau Interpersonal Relations based IPSRT will be applied to the intervention group, and the control group will be given a CMHS and will also continue the treatment. IPSRT will take 40-45 minutes twice in a week and will be conducted in 10-12 individual meetings in total. Immediately, 1 month and 3 months after the interviews, post-tests will be applied to the intervention and control groups With this study, the biological rhythms of IPSRT individuals based on Peplau Interpersonal Relationship Theory in bipolar disorder will be regulated and the frequency of relapse will decrease. In addition, individuals with bipolar disorder, which is one of the lifelong mental illnesses that cause stigmatization, will continue their lives in the community, their functionality will increase in their work life, school life and social life, and hospitalization will decrease

DETAILED DESCRIPTION:
Interpersonal and Social Rhythm Therapy (IPSRT) is a type of psychotherapy that applies social rhythm theories in bipolar disorder. The purpose of IPSRT is to stabilize people's social routines (daily routines, sleep-wake balances), gain insight into the two-way relationship between interpersonal events and mood, and increase their satisfaction with social roles.The main purpose is to increase functionality in bipolar disorder. Using this versatile approach, IPSRT aims to improve current mood and teach patients skills to protect themselves against the development of new bipolar episodes. In individuals with bipolar disorder; Non-compliance with pharmacological treatment, stressful life events and disturbances in social rhythms cause relapses. As a component of KIPT-SRT is psychoeducation, education about the disease and treatment is provided to ensure compliance with pharmacological treatment IPSRT seeks to reduce patients' interpersonal and social-based stress factors by addressing interpersonal and social role problems. It also increases the stability of social rhythms by organizing daily routines, paying attention to the extent to which positive and negative life events can affect these daily routines Psychiatric nursing is an interpersonal process in which a professional nurse helps to improve the mental health of the individual, family and society, to prevent mental illness and suffering experiences or to cope with the disease and, if necessary, to find meaning from these experiences (Kum,1996; Çam, 2014). Peplau, one of the psychiatric nursing theorists, believed that many nursing problems arise from human relationships, and nursing interventions should be planned in this direction in order for individuals to continue their development and to solve these problems. The interpersonal process is at the center of the model, as nurses can recognize and help solve problems arising from human relationships. Interview steps of IPSRT, which has features that overlap with Peplau's theory of interpersonal relations, are seen to be parallel with Peplau's relationship steps between nurse and patient. On the basis of this theory, the application of IPSRT can be used as an important strategy by psychiatric nurses in reducing the frequency of recurrence in bipolar disorder patients who continue to experience bipolar attacks. This study will be carried out in order to evaluate the difference in terms of biological rhythm and recurrence frequency between the intervention and control group of IPSRT based on Peplau's theory of Interpersonal Relationships This study was planned as a follow-up study in a quantitative, randomized controlled experimental design, aiming to determine the effectiveness of Peplau's Interpersonal Relations theory-based IPSRT applied to individuals with bipolar disorder to determine the effect on biological rhythm, interpersonal relationships and relapse frequencies. Pre-intervention pre-test, post-intervention post-test and follow-up scheme will be used. To carrying out of this study, first of all, intervention and control groups will be formed by randomization according to gender and bipolar type (I-II), using the Introductory Information Form, Young Mania Rating and Hamilton Depression Rating Scales from individuals with bipolar disorder registered to the Community Mental Health Service (CMHS). As a pre-test (Introductory Information Form, Young Mania Rating Scale, Hamilton Depression Rating Scale, Biological Rhythm Assessment Interview, Interpersonal Competence Scale) to the intervention and control groups, Peplau Interpersonal Relations based IPSRT will be applied to the intervention group, and the control group will be given a CMHS and will also continue the treatment. IPSRT will take 40-45 minutes twice in a week and will be conducted in 10-12 individual meetings in total. Immediately, 1 month and 3 months after the interviews, post-tests will be applied to the intervention and control groups.

With this study, the biological rhythms of IPSRT individuals based on Peplau Interpersonal Relationship Theory in bipolar disorder will be regulated and the frequency of relapse will decrease. In addition, individuals with bipolar disorder, which is one of the lifelong mental illnesses that cause stigmatization, will continue their lives in the community, their functionality will increase in their work life, school life and social life, and hospitalization will decrease

ELIGIBILITY:
Inclusion Criteria:

* Adult individuals with bipolar disorder according to DSM-V diagnostic criteria
* Those who agreed to participate in the research
* Those who are at a level that can understand scales and forms with the competence to carry out individual interviews
* Individuals who are open to communication and cooperation and have no language problems

Exclusion Criteria:

* Individuals with psychotic findings,
* Individuals with a diagnosis of schizoaffective.
* Those who want to quit their job and leave
* Those who cannot adapt, those who have communication problems
* Those who did not attend at least 3 interviews of IPT-SRT
* 12 points or higher from the Young Mania Rating Scale
* A score of 18 or higher on the Hamilton Depression Scale

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Young Mania rating scale scores | about 3 months
  Change from baseline in Young Mania rating scale scores at 3 months
Biological Rhythm Interview Evaluation scores | about 3 months
  Change in Biological Rhythm Interview Evaluation scores in 3 months compared to baseline
Hamilton Depression rating scale scores | about 3 months
  Change from baseline in Hamilton Depression rating scale scores at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Şeyda Dülgerler, Principal Investigator — Ege University Nursing
Locations (1):
- İzmir Katip Çelebi University Atatürk Eğitim ve Araştırma Hastanesi, Izmir, Karabağlar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Goldstein TR, Fersch-Podrat R, Axelson DA, Gilbert A, Hlastala SA, Birmaher B, Frank E. Early intervention for adolescents at high risk for the development of bipolar disorder: pilot study of Interpersonal and Social Rhythm Therapy (IPSRT). Psychotherapy (Chic). 2014 Mar;51(1):180-9. doi: 10.1037/a0034396. Epub 2013 Dec 30. PMID 24377402
- [Result] Crowe M, Inder M, Douglas K, Carlyle D, Wells H, Jordan J, Lacey C, Mulder R, Beaglehole B, Porter R. Interpersonal and Social Rhythm Therapy for Patients With Major Depressive Disorder. Am J Psychother. 2020 Mar 1;73(1):29-34. doi: 10.1176/appi.psychotherapy.20190024. Epub 2019 Nov 22. PMID 31752508
- [Result] Mizushima H. [Psychoeducation and interpersonal and social rhythm therapy for bipolar disorder]. Seishin Shinkeigaku Zasshi. 2011;113(9):880-5. Japanese. PMID 22117393
- [Result] Crowe M, Porter R, Inder M, Carlyle D, Luty S, Lacey C, Frampton C. Clinical Effectiveness Trial of Adjunctive Interpersonal and Social Rhythm Therapy for Patients With Bipolar Disorder. Am J Psychother. 2020 Sep 1;73(3):107-114. doi: 10.1176/appi.psychotherapy.20190035. Epub 2020 Apr 20. PMID 32306747

DOCUMENTS (2):
  • Study Protocol (2022-05-15): https://cdn.clinicaltrials.gov/large-docs/92/NCT05420792/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-15): https://cdn.clinicaltrials.gov/large-docs/92/NCT05420792/SAP_001.pdf